CLINICAL TRIAL: NCT02448225
Title: PET Imaging of Lung Cancer and Indeterminate Pulmonary Nodules With 18F-FSPG
Brief Title: 18F-FSPG PET/CT in Imaging Patients With Newly Diagnosed Lung Cancer or Indeterminate Pulmonary Nodules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Chirayu Shah, Associate Professor of Clinical Radiology, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC THO 1524; NCI-2015-00748 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA068485 (NIH)
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Results first posted 2022-05-10 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Lung Carcinoma; Solitary Pulmonary Nodule; Cigarette Smoking Behavior
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule; Cigarette Smoking | interventions — Fluorodeoxyglucose F18; 4-(3-fluoropropyl)glutamic acid; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (18F-FDG PET/CT, 18F-FSPG PET/CT) (Experimental): Patients undergo 18F-FDG PET/CT scan per standard of care. Within 15 working days, patients also undergo 18F-FSPG PET scan over 60 minutes followed by an 18F-FSPG PET/CT scan over 30 minutes.
  Interventions: Procedure: Computed Tomography; Radiation: fluorodeoxyglucose F-18; Drug: Fluorine F 18 L-glutamate Derivative BAY94-9392; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography; Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Procedure: Computed Tomography — Undergo 18F-FDG PET/CT - standard of care
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Procedure: Computed Tomography — Undergo 18F-FSPG PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Radiation: fluorodeoxyglucose F-18 — Undergo 18F-FDG PET/CT - standard of care
  Other Names: 18FDG; FDG; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose
Drug: Fluorine F 18 L-glutamate Derivative BAY94-9392 — Undergo 18F-FSPG PET/CT
  Other Names: (S)-4-(3-18F-fluoropropyl)-L-glutamic Acid; 18F-FSPG; BAY94-9392
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo 18F-FDG PET/CT - standard of care
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; proton magnetic resonance spectroscopic imaging
Procedure: Positron Emission Tomography (PET) — Undergo 18F-FSPG PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; Positron Emission Tomography Scan; proton magnetic resonance spectroscopic imaging

SUMMARY:
This clinical trial compares fluorine F 18 L-glutamate derivative BAY94-9392 (18F-FSPG) positron emission tomography (PET)/computed tomography (CT) to the standard of care fluorodeoxyglucose F-18 (18F-FDG) PET/CT in imaging patients with newly diagnosed lung cancer or indeterminate pulmonary nodules. PET/CT uses a radioactive glutamate (one of the common building blocks of protein) called 18F-FSPG which may be able to recognize differences between tumor and healthy tissue. Since tumor cells are growing, they need to make protein, and other building blocks, for cell growth that are made from glutamate and other molecules. PET/CT using a radioactive glutamate may be a more effective method of diagnosing lung cancer than the standard PET/CT using a radioactive glucose (sugar), such as 18F-FDG.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the imaging characteristics of 18F-FSPG PET/CT with standard-of-care, 18F-FDG PET/CT.

II. To compare the imaging characteristics of 18F-FSPG PET/CT to standard-of-care 18F-FDG PET/CT in patients with newly diagnosed lung cancer.

III. To determine whether 18F-FSPG uptake in lung cancer can be predicted based on correlation with CD44 and amino acid transport system xc- (xC-) expression in surgical pathology specimens.

OUTLINE:

Patients undergo 18F-FDG PET/CT scan per standard of care. Within 15 working days, patients also undergo 18F-FSPG PET scan over 60 minutes followed by an 18F-FSPG PET/CT scan over 30 minutes.

After completion of study, patients are followed up for 2 years if needed for diagnosis.

ELIGIBILITY:
Inclusion Criteria:

- Have an indeterminate untreated pulmonary nodule (IPN) (7-30 mm diameter) on CT, or an indeterminate lung mass (> 30 mm diameter), without prior examinations that establish that the lesion has been stable for two or more years, untreated.

or

* Have a newly diagnosed, untreated primary lung cancer diameter 7 mm or more.
* Be able to give informed consent, which will include a layman's explanation of the estimated amount of additional radiation that the patient will receive from the investigational PET/CT scan using 18F-FSPG
* Must agree at the time of study entry to undergo clinically indicated biopsy(ies) or a 24-month period of follow-up, as needed, to resolve the etiology of their IPN(s) or lung mass(es).

Exclusion Criteria:

* Pregnant or lactating patients will be excluded, as will females of childbearing potential who refuse to undergo a serum or urinary beta-HCG pregnancy test the day of either the 18F-FSPG or the 18F-FDG PET/CT scans, in accordance with the standard policy of the Medical Imaging Service at our facility. Women who have experienced 24 consecutive months of amenorrhea, have reached at least 60 years of age, or have had a tubal ligation or hysterectomy documented in their medical records are considered not to be of childbearing potential for the purposes of this protocol
* Patients with a body weight of 400 pounds or more or a body habitus or disability that will not permit the imaging protocol to be performed
* A recognized active lung infection
* Previous systemic or radiation treatment for cancer of any type within 1 year
* For patients who do not have a tissue diagnosis:

  * Non-oncologic severe co-morbidities suggesting a life span of less than two years if not treated, as determined by the potential subject's treating physician.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2022-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chirayu Shah, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Tennessee Valley Health System Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 46 patients between two clinical sites (15 at Veterans Affairs-Tennessee Valley Health System Nashville, TN and 31 at Vanderbilt University Medical Center, Nashville, TN). The enrollment period was 6/16/15 to 1/5/21.
Period: Overall Study
Arm/Group | Diagnostic (18F-FDG PET/CT, 18F-FSPG PET/CT)
Started | 46
Completed | 26
Not Completed | 20
Not completed — Withdrawal by Subject | 1
Not completed — Did not get FSPG scan | 18
Not completed — Treated between the FDG and FSPG scan | 1

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (18F-FDG PET/CT, 18F-FSPG PET/CT)
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Ability of 18F-FSPG PET/CT to Discriminate Benign From Malignant Nodules
Description: Sensitivity, specificity, overall accuracy and receiver operating characteristic (ROC) curves will be generated and compared for both 18F-FDG and 18F-FSPG tests.
  Sensitivity is the proportion of High(positive) among cancer patients. Specificity is the proportion of low(negative) among benign tumors. Accuracy is the proportion of correctly diagnosed among analyzed patients. Area under the curve(AUC) is the area under the ROC curve, which is the plot of sensitivity by 1-specificity.
Time Frame: Up to 2 years
Population: Patients analyzed among enrolled patients
Measure: Number (95% Confidence Interval); unit: proportion, range 0 to 1, higher better
Arm/Group | Diagnostic (18F-FDG PET/CT, 18F-FSPG PET/CT)
Number analyzed (Participants) | 26
proportion, range 0 to 1, higher better
  FDG sensitivity(low and high) | 0.706 [0.489 to 0.922]
  FDG specificity | 0.778 [0.506 to 1.000]
  FDG accuracy | 0.731 [0.560 to 0.901]
  FDG AUC(area under curve) | 0.817 [0.653 to 0.981]
  ESPG sensitivity(low and high) | 0.824 [0.642 to 1.000]
  ESPG specificity(low and high) | 0.667 [0.359 to 0.975]
  ESPG accuracy | 0.769 [0.607 to 0.931]
  ESPG AUC | 0.843 [0.682 to 1.000]

2. Secondary Outcome: CD44 and xC- Expression Levels in Tissue Samples(0-3)
Description: The level of expression of xCT and CD44 proteins in the cytoplasmic membrane of tumor cells were examined by an experienced pathologist who was blinded to any patient and imaging information. The percentage of tumor cells positive for the marker and the intensity of staining were evaluated, the latter using a scale of 0 (none), 1+ (weak), 2+ (intermediate), and 3+ (strong) with a sample being reported as positive if greater than 10% of the tumor cells in the sample were positively stained with any intensity.
Time Frame: Up to 2 years
Population: 12 cancer patients among those enrolled.
Measure: Mean (Standard Deviation); unit: IHC score, range 0 and above
Groups:
- Some Cancer Patients: Patients undergo 18F-FDG PET/CT scan per standard of care. Within 15 working days, patients also undergo 18F-FSPG PET scan over 60 minutes followed by an 18F-FSPG PET/CT scan over 30 minutes.
  Computed Tomography: Undergo 18F-FDG PET/CT - standard of care
  Computed Tomography: Undergo 18F-FSPG PET/CT
  fluorodeoxyglucose F-18: Undergo 18F-FDG PET/CT - standard of care
  Fluorine F 18 L-glutamate Derivative BAY94-9392: Undergo 18F-FSPG PET/CT
  Laboratory Biomarker Analysis: Correlative studies
  Positron Emission Tomography: Undergo 18F-FDG PET/CT - standard of care
  Positron Emission Tomography (PET): Undergo 18F-FSPG PET/CT
Arm/Group | Some Cancer Patients
Number analyzed (Participants) | 12
IHC score, range 0 and above
  CD44 | 2.6 (0.5)
  xCT | 1 (1)

3. Secondary Outcome: Uptake of 18F-FSPG (Expressed in Maximal Standardized Uptake Value [SUV] Within the Tumor)
Description: Maximum standardized uptake values (SUVmax) were normalized to lean body mass and measured with a 1 cm diameter round region of interest over the area of greatest uptake in the lesion being measured.
Time Frame: Up to 2 years
Population: enrolled patients included 7 benign and 19 cancer patients.
Measure: Mean (Standard Deviation); unit: Maximum standardized uptake values (SUVm
Groups:
- Benign Patients: Patients undergo 18F-FDG PET/CT scan per standard of care. Within 15 working days, patients also undergo 18F-FSPG PET scan over 60 minutes followed by an 18F-FSPG PET/CT scan over 30 minutes.
  Computed Tomography: Undergo 18F-FDG PET/CT - standard of care
  Computed Tomography: Undergo 18F-FSPG PET/CT
  fluorodeoxyglucose F-18: Undergo 18F-FDG PET/CT - standard of care
  Fluorine F 18 L-glutamate Derivative BAY94-9392: Undergo 18F-FSPG PET/CT
  Laboratory Biomarker Analysis: Correlative studies
  Positron Emission Tomography: Undergo 18F-FDG PET/CT - standard of care
  Positron Emission Tomography (PET): Undergo 18F-FSPG PET/CT
- Cancer Patients: Patients undergo 18F-FDG PET/CT scan per standard of care. Within 15 working days, patients also undergo 18F-FSPG PET scan over 60 minutes followed by an 18F-FSPG PET/CT scan over 30 minutes.
  Computed Tomography: Undergo 18F-FDG PET/CT - standard of care
  Computed Tomography: Undergo 18F-FSPG PET/CT
  fluorodeoxyglucose F-18: Undergo 18F-FDG PET/CT - standard of care
  Fluorine F 18 L-glutamate Derivative BAY94-9392: Undergo 18F-FSPG PET/CT
Arm/Group | Benign Patients | Cancer Patients
Number analyzed (Participants) | 9 | 17
Maximum standardized uptake values (SUVm | 0.8 (0.7) | 3.9 (3.6)

4. Secondary Outcome: Ability of 18F-FSPG PET/CT to Stage of Lung Cancer (Metastatic or Not)
Description: Sensitivity, specificity, overall accuracy and ROC curves will be generated and compared for both 18F-FDG and 18F-FSPG tests. Wilcoxon rank-sum or Kruskal-Wallis tests will be applied for the group comparisons of the biodistribution characteristics of 18F-FDG and 18F-FSPG tests.
  Sensitivity is the proportion of High(positive) among cancer patients. Specificity is the proportion of low(negative) among benign tumors. Accuracy is the proportion of correctly diagnosed among all patients. Area under the curve(AUC) is the area under the ROC curve.
Time Frame: Up to 2 years
Population: Cancer patients enrolled.
Measure: Number (95% Confidence Interval); unit: proportion, range 0-1, higher better
Arm/Group | Diagnostic (18F-FDG PET/CT, 18F-FSPG PET/CT)
Number analyzed (Participants) | 17
proportion, range 0-1, higher better
  FDG sensitivity | 0.8 [0.552 to 1]
  FDG specificity | 0.857 [0.598 to 1]
  FDG accuracy | 0.824 [0.642 to 1]
  FDG AUC | 0.871 [0.7 to 1]
  FSPG sensitivity | 0.2 [0 to 0.448]
  FSPG specificity | 0.286 [0 to 0.62]
  FSPG accuracy | 0.235 [0.034 to 0.437]
  FSPG AUC | 0.8 [0.594 to 1]

5. Other Pre Specified Outcome: Uptake of 18F-FSPG (Expressed in Maximal Standardized Uptake Value [SUV] Within the
Description: Descriptive statistics, including means, standard deviations, and ranges for continuous
Time Frame: Up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From study entry to approximately 60 days
Arm/Group | Diagnostic (18F-FDG PET/CT, 18F-FSPG PET/CT)
All-Cause Mortality (participants affected / at risk) | 6/46
Serious Adverse Events (participants affected / at risk) | 1/46
Other Adverse Events (participants affected / at risk) | 7/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (18F-FDG PET/CT, 18F-FSPG PET/CT) (N=46)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (18F-FDG PET/CT, 18F-FSPG PET/CT) (N=46)
Non-cardiac chest pain (General disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT02448225/Prot_SAP_000.pdf